CLINICAL TRIAL: NCT00382083
Title: Premedication to Reduce Discomfort With Screening Mammography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mountain States Tumor and Medical Research Institute (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MSTMRI - 001
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2006-09-28 (Estimated); Status verified 2006-09

CONDITIONS: Breast Pain
Keywords: Mammogram; Pain; Discomfort; Breast; Pre-medication
MeSH Terms: conditions — Mastodynia; Pain | interventions — Acetaminophen; Ibuprofen

INTERVENTIONS:
Drug: 1000 mg acetaminophen
Drug: 800 mg ibuprofen
Drug: 1 oz 4% lidocaine gel

SUMMARY:
This study will explore the effect of pre-medication with acetaminophen, ibuprofen, and topical lidocaine gel (Topicaine) on the perception of discomfort and overall satisfaction with the mammography experience.

The research questions are:

1. What is the relationship between the use of acetaminophen, ibuprofen, and Topicaine prior to screening mammography and the perception of discomfort during the procedure?
2. What is the relationship between perception of discomfort and overall satisfaction with the mammography experience?
3. What is the relationship between the perception of discomfort and plans for future mammograms?
4. What other factors are associated with the perception of discomfort and satisfaction?

DETAILED DESCRIPTION:
Breast cancer is prevalent, deadly, costly, and has low cure rates unless detected in its early stages. Mammography is the key component to early detection, yet it remains underutilized due to cost, access, and factors such as fear of pain.

Multiple studies have shown that most women find mammography uncomfortable, even painful. Yet, little research has been done to find methods to reduce mammography-related discomfort. In an unpublished Master's thesis, this investigator found that women who expected discomfort > 40 on a visual analog scale (VAS) who were pre-medicated with 1000 mg of acetaminophen reported lower discomfort scores than those pre-medicated with placebo, but the sample size was too small to reach statistical significance. Further study on the effects of pre-medication is needed.

Pain should not be associated with a potentially lifesaving procedure. A more comfortable and positive experience with mammography may increase the number of women who participate in regular mammography screening, and, thereby, increase early detection and reduce the mortality rate, costs, and emotional trauma associated with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for age-appropriate screening mammography at St. Luke's Breast Cancer Detection Center
* Expect discomfort of 40 or greater on a scale of 0-100
* Willing to arrive 1 hour early for appointment to enroll in study

Exclusion Criteria:

Women who:

* expect discomfort from their mammogram to be < 40 on a scale of 0-100
* cannot understand or read English or who are unable to complete the consent process or questionnaire for reasons such as hearing impairment or other physical or mental disabilities
* have a sensitivity or allergy to acetaminophen, ibuprofen, or lidocaine
* have significant liver or kidney dysfunction
* are breast-feeding
* cannot arrive a minimum of 60 minutes earlier than their appointment time
* have taken any pain relief medications within 24 hours of their mammogram appointment, including over-the-counter medications.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-03; Study Completion 2006-06

PRIMARY OUTCOMES:
Discomfort scores on a visual analog scale at recruitment, at enrollment, and after mammogram
Satisfaction scores on a visual analog scale after mammogram

SECONDARY OUTCOMES:
Pre-mammogram anxiety scores on a visual anxiety scale at enrollment
Pre-mammogram breast tenderness scores on a visual analog scale at enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Colleen K. Lambertz, MSN, FNP, Principal Investigator — Mountain States Oncology Group; Paul G Montgomery, MD, Study Chair — St. Luke's Mountain States Tumor Institute; Theodore A Walters, MD, Study Director — Mountain States Tumor Medical Research Institute
Locations (1):
- St. Luke's Mountain States Tumor Institute Breast Cancer Detection Center, Boise, Idaho, United States